CLINICAL TRIAL: NCT00625352
Title: Prospective Phase II Trial of a Combination of Gemcitabine and UFT as First-Line Treatment in Elderly Patients With Advanced Non-Small Cell Carcinoma
Brief Title: Study of Developing an Optimal Gemcitabine Based Regimen to Treat Elderly Patients With Advanced Non-Small Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ulsan University Hospital (Other)
Collaborators: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Young Joo Min/Associate professor, Ulsan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UUH-ONC-0019
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2008-02-28 (Estimated); Status verified 2008-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Carcinoma, Non-Small-Cell Lung; Aged; Gemcitabine; UFT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Tegafur

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Gemcitabine, UFT — Gemcitabine 1,250mg/m2 IV on D1 and D8 of every 3 weeks combined with UFT 400mg daily PO for 14 days every 3 weeks. Gemcitabine will be administered to patients a maximum of 4 cycles, and then discontinued. UFT will be continued until progression.

SUMMARY:
Cares for elderly patients with advanced non-small cell lung cancer(NSCLC) become one of the common clinical practices oncologist are now facing. So, we need to seek adequate regimens for them. Gemcitabine is well known to be one of active third generation agents in terms of both efficacy and tolerability. Gemcitabine alone have been recommended as first line treatment for elderly NSCLC patients, especially in the aspect of tolerability. However, gemcitabine alone is suggested to be suboptimal to control their disease. Therefore, we plan to make an optimal regimen containing gemcitabine for the elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically- confirmed Non-Small-Cell Lung Cancer Stage IIIB/IV
* No prior chemotherapy
* Existence of measurable disease. The measurable disease should not have been irradiated
* Life expectancy of more than 3 months
* Age ≥ 70 years
* Performance status (ECOG):1 or 2
* Adequate bone marrow function (Absolute neutrophil count >1500/mm^3, Platelet count>100000/mm^3, Hemoglobin>9gr/mm^3)
* Adequate liver (Bilirubin<2 times upper limit of normal and SGOT/SGPT<3 times upper limit of normal) and renal function (creatinine<1.5mg/dl)
* Informed consent

Exclusion Criteria:

* Psychiatric illness or social situation that would preclude study compliance.
* Other concurrent uncontrolled illness.
* Other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* Currently/recently taken warfarin, phenprocoumon or phenytoin
* Hypersensitivity history to any drug

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
overall response rate | every two cycles

SECONDARY OUTCOMES:
toxicity, response duration, progression free survival, overall survival | according to protocol

CONTACTS AND LOCATIONS:
Locations (1):
- Ulsan University Hospital, Ulsan, South Korea